CLINICAL TRIAL: NCT02075736
Title: The Effect of KTP (Potassium-titanyl-phosphate) Green Light Prostatectomy (120W) Compared With TUR-P When Treating Benign Prostatic Hyperplasia in High Risk Patients, A Prospective Randomized Study
Brief Title: KTP Green Light Prostatectomy Compared With TUR-P in High Risk Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Hannu Koistinen, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35/13/03/02/08
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KTP laser (Experimental): device
  Interventions: Procedure: KTP laser
- TUR-P (Active Comparator): device
  Interventions: Procedure: TUR-P

INTERVENTIONS:
Procedure: KTP laser
  Other Names: Green laser
  Arms: KTP laser
Procedure: TUR-P — device
  Arms: TUR-P

SUMMARY:
The purpose of this study is to compare safety and efficacy of Green Light PVP (Photoselective Vaporization of the Prostate) compared to TUR-P in high risk patients

ELIGIBILITY:
Inclusion Criteria:

* Men with anticoagulant medication undergoing surgery for BPH

Exclusion Criteria:

* Previous prostate surgery
* Carcinoma of the prostate
* Neurogenic bladder
* Bladder carcinoma

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-bleeding rate requiring hospitalization | two months postoperatively

SECONDARY OUTCOMES:
IPSS (International Prostate Symptom Score) | 0, 3, 6 and 12 months
  symptom score
DAN-PSS (Danish Prostate Symptom Score) | 0, 3, 6 and 12 months
Maximum flow rate (Qmax) | 0, 3, 6 and 12 months
Residual urine | 0, 3, 6 and 12 months
Length of catheterization | Participants will be followed for the duration of hospital stay, an expected maximum of one week
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected maximum of one week
Perioperative bleeding | Time of operation
IIEF (International Index of Erectile Function) questionnaire | 0,12 months
TRUS (transrectal ultrasound) | 0, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland